CLINICAL TRIAL: NCT02827630
Title: Use of Proteus Discover to Enable Improved Clinical Outcomes in Subjects With Uncontrolled Hypertension and Type 2 Diabetes Mellitus: A Pilot Study
Brief Title: Proteus Discover in Subjects With Uncontrolled Hypertension and Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Proteus Digital Health, Inc. (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PB-DISC_CMB_01
Record Dates: First submitted 2016-06-29; First posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Hypertension; Diabetes Mellitus, Type 2; Hypercholesterolemia
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2; Hypercholesterolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- DH-4 (Active Comparator): Subjects will use Proteus Discover, the digital health offering (DH) for 4 weeks
  Interventions: Other: Proteus Discover
- DH-12 (Active Comparator): Subjects will use Proteus Discover, the digital health offering (DH) for 12 weeks
  Interventions: Other: Proteus Discover
- Usual Care (Other): Subjects received usual medical care including all normal interventions such as medication titration, adherence counseling, lifestyle coaching, and additional clinic visits per their providers' discretion.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Proteus Discover — FDA cleared Wearable Sensor with Ingestible Sensor and Mobile Device Application
  Arms: DH-12; DH-4
Other: Usual Care — Routine medical care including medication titration, adherence counseling, and lifestyle coaching.
  Arms: Usual Care

SUMMARY:
The purpose of this study was to evaluate the efficacy of a new digital health offering, Proteus Discover to lower blood pressure and glycated hemoglobin in patients with uncontrolled hypertension and type 2 diabetes.

DETAILED DESCRIPTION:
"Cardiometabolic diseases" as defined in this protocol refer to diseases that increase risk for cardiovascular disease. Proteus® Digital Health is operationally defining cardiometabolic (CMB) conditions for this study as including hypertension, type 2 diabetes, and hypercholesterolemia. The prevalence of metabolic diseases is growing. Factors contributing to this rise include the obesity epidemic and the aging population. In particular, because of the costs and risk of complications associated with diabetes and hypertension, many health systems and payers are increasing focus on interventions to reduce the burden of these diseases.

The purpose of the study was to evaluate the ability of a new digital health offering, Proteus Discover to lower blood pressure and glycated hemoglobin in patients with uncontrolled hypertension and type 2 diabetes.

The study enrolled subjects with uncontrolled hypertension and type 2 diabetes failing at least 2 antihypertensives and metformin and/or a sulfonylurea. Subjects were randomized to one of 3 arms: use of Proteus Discover for 4 weeks, use of Proteus Discover for 12 weeks, or usual care.

Subjects randomized to the intervention arms, used a digital health offering to (1) provide automatic and passive electronic documentation of medication adherence and patterns of medication taking, (2) assist providers in distinguishing inadequate medication adherence or pharmacologic unresponsiveness as the root cause for uncontrolled hypertension and type 2 diabetes, and (3) inform management decisions (dose adjustment, medication addition or substitution, adherence counseling, referral to a hypertension specialist).

Subjects randomized to usual care, received usual medical care such as medication changes, adherence counseling, and lifestyle coaching. Providers could also schedule additional visits without restrictions.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 to 75 years old) who are diagnosed with essential hypertension and type 2 diabetes mellitus with or without hypercholesterolemia (defined as taking statin therapy).
* Both hypertension and diabetes are suboptimally controlled at Screening:

  1. SBP is ≥ 140 mm Hg (and his/her BP goal is < 140/90 mm Hg).
  2. A1C is ≥ 7% and ≤ 11% at Screening (A1C is above goal by ≥ 0.5%).
* On a stable anti-hypertensive regimen (on current regimen for at least 30 days) with at least 2 anti-hypertensive medications
* Ability to manage the subject during the 12-week study with anti-hypertensive medication(s) and dose forms (or same drug classes and comparable doses for Usual Care subjects) used within the study.
* Currently on metformin and/or glipizide for diabetes for at least the past 60 days prior to Screening. Subjects can be managed on other noninsulin diabetes medicines (including sulfonylureas other than glipizide) during the study.
* Subjects must have a Proteus test pill (IS used to test that the Proteus Patch is correctly placed on the body and paired with the mobile device) detected as part of onboarding on the Proteus device (during the Proteus Onboarding Visit).
* In the Investigator's opinion inadequate medication adherence is a potential factor in the subject's uncontrolled hypertension or diabetes.

Exclusion Criteria:

* BMI > 40 kg/m2 as subjects may be more likely to have secondary reasons for out of control blood pressure (BP) and/or diabetes.
* History of skin sensitivity to adhesive medical tape or metals for subjects in the Intervention Arms.
* History of acute or chronic dermatitis for subjects in the Intervention Arms.
* Any condition that in the investigator's opinion could preclude safe participation in the study.
* Secondary cause for hypertension (eg, renal impairment or renal artery stenosis) or uncontrolled diabetes (eg, corticosteroid use).
* Mean SBP ≥ 180 mm Hg and/or DBP ≥ 110 mm Hg, if associated with evidence of hypertensive emergency..
* Current or recent (within past year) treatment with insulin or other injectables for diabetes.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2015-05; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Week 4 Change in Systolic Blood Pressure | 4 weeks

SECONDARY OUTCOMES:
Change in Diastolic Blood Pressure | 4 weeks
Proportion at blood pressure goal | 4 weeks
  BP < 140/90 mmHg
Proportion at blood pressure goal | 12 weeks
  BP < 140/90 mmHg
Change in Systolic Blood Pressure | 12 weeks
Change in Diastolic Blood Pressure | 12 weeks
Change in fasting plasma glucose | 4 weeks
Change in fasting plasma glucose | 12 weeks
Change in glycated hemoglobin | 12 weeks
Average Daily Medication Adherence as Measured by DH | 4 weeks
  Medication adherence by medication and overall (aggregate average of daily adherence to each of the medications) in all DH subjects. Reported as a %.
Average Daily Medication Adherence as Measured by DH | 4 to 12 weeks
  Medication adherence by medication and overall (aggregate average of daily adherence to each of the medications) DH-12 subjects. Reported as a %.
Average daily physical activity duration as measured by DH in DH-12 subjects | 4 to 12 weeks
Average daily rest duration as measured by DH in DH-12 subjects | 4 to 12 weeks
Average daily step count as measured by DH in DH-12 subjects | 4 to 12 weeks
Average daily step count as measured by DH in all DH subjects | 4 weeks
Average daily physical activity duration as measured by DH in all DH subjects | 4 weeks
Average daily rest duration as measured by DH in all DH subjects | 4 weeks
Table Summary of the Number of Subjects with Medication Changes | 4 weeks
  Summary table of the number of medication dose increases, medication dose decreases, medication stops, medication additions, and no change. Data was summarized separately for hypertension, type 2 diabetes, and hypercholesterolemia. Data to be collected on CRF. Data summarized by type of medication change.
Table Summary of the Number of Subjects with Medication Changes | 12 weeks
  Summary table of the number of medication dose increases, medication dose decreases, medication stops, medication additions, and no change. Data was summarized separately for hypertension, type 2 diabetes, and hypercholesterolemia. Data to be collected on CRF. Data summarized by type of medication change.
Table Summary of the Number of Subjects with Medical Decisions Other than Medication Changes | 2 weeks
  Number of subjects who received adherence counseling, patient education, referral to a specialist, referral to disease management, lifestyle changes, and other medical decisions. Data summarized by type of decision.
Table Summary of the Number of Subjects with Medical Decisions Other than Medication Changes | 4 weeks
  Number of subjects who received adherence counseling, patient education, referral to a specialist, referral to disease management, lifestyle changes, and other medical decisions. Data summarized by type of decision.
Table Summary of the Number of Subjects with Medical Decisions Other than Medication Changes | 12 weeks
  Number of subjects who received adherence counseling, patient education, referral to a specialist, referral to disease management, lifestyle changes, and other medical decisions. Data summarized by type of decision.
Number of Treatment-Related Adverse Events | 12 weeks
  Descriptive summary of adverse events for DH arms versus usual care

OTHER OUTCOMES:
Change in LDL in subjects using a statin | 4 weeks
Change in LDL in subjects using a statin | 12 weeks
Change in ACC/AHA ASCVD 10-year risk | 4 weeks
Change in ACC/AHA ASCVD 10-year risk | 12 weeks
  American College of Cardiology/ American Heart Association Atherosclerotic Cardiovascular Disease Risk Score
Change in Patient Activation Measure (PAM) | 4 weeks
  PAM is a validated measure of patient activation
Change in Patient Activation Measure (PAM) | 12 weeks
  PAM is a validated measure of patient activation
Resource Utilization: Summary of the number of outpatient visits, ER visits, and hospitalizations during the study | 12 weeks
  Data to be summarized descriptively
Proportion of subjects with adequate activity and rest information while using Proteus Discover | 4 weeks
Proportion of subjects with adequate activity and rest information while using Proteus Discover | 12 weeks
Change in weight in kg | 4 weeks
Change in weight in kg | 12 weeks
Change in BMI in kg/m^2 | 4 weeks
Change in BMI in kg/m^2 | 12 weeks
Change in waist circumference (cm) | 4 weeks
Change in waist circumference (cm) | 12 weeks
Subject Reported Outcomes: Results from a subject satisfaction [to DH] questionnaire administered at the end of using DH. | 4 or 12 weeks
  Satisfaction (with Proteus Discover) survey administered upon completion of use of Proteus Discover
Provider Reported Outcomes: Results from a provider satisfaction [to DH] questionnaire administered at the end of using DH. | 4 or 12 weeks
  Satisfaction (with Proteus Discover) survey administered upon completion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Lars Osterberg, MD, Principal Investigator — Stanford University

REFERENCES:
- [Background] Centers for Disease Control and Prevention (CDC). Vital signs: prevalence, treatment, and control of high levels of low-density lipoprotein cholesterol--United States, 1999-2002 and 2005-200. MMWR Morb Mortal Wkly Rep. 2011 Feb 4;60(4):109-14. PMID 21293326
- [Derived] Frias J, Virdi N, Raja P, Kim Y, Savage G, Osterberg L. Effectiveness of Digital Medicines to Improve Clinical Outcomes in Patients with Uncontrolled Hypertension and Type 2 Diabetes: Prospective, Open-Label, Cluster-Randomized Pilot Clinical Trial. J Med Internet Res. 2017 Jul 11;19(7):e246. doi: 10.2196/jmir.7833. PMID 28698169
- See also: American Diabetes Association. Statistics about diabetes. — http://www.diabetes.org/diabetes-basics/statistics/?loc=db-slabnav